CLINICAL TRIAL: NCT00547534
Title: Pilot Study of Bortezomib, Bendamustine and Rituximab for Patients With Relapsed or Refractory, Indolent or Mantle Cell Non-Hodgkin's Lymphoma
Brief Title: Pilot Study of Bortezomib, Bendamustine and Rituximab on Non-Hodgkin's Lymphoma
Acronym: BVR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Cephalon (Industry)
Responsible Party: Principal Investigator, Jonathan Friedberg, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULYM07054
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-07

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Bortezomib; Bendamustine; Rituximab; Relapsed; Refractory; Mantle Cell; Indolent
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Bortezomib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lymphoma Subjects receiving protocol therapy (Experimental): Subjects that met all eligibility criteria and were treated with Bendamustine, Rituxan and Bortezomib.
  Interventions: Drug: bortezomib; Drug: bendamustine; Drug: rituximab

INTERVENTIONS:
Drug: bortezomib — 1.3 mg/m^2 on days 1, 4, 8, 11
  Other Names: Velcade
Drug: bendamustine — 90 mg/m^2 days 1 and 4
  Other Names: Treanda
Drug: rituximab — 375 mg/m^2 day 1
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to evaluate how non-Hodgkin's lymphoma that has not responded to, or that has returned after standard treatment, responds to bortezomib, rituximab and bendamustine, and also to see what effects this drug combination have on this cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-specific procedure not part of routine medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use acceptable method of birth control for duration of study.
* Male subject agrees to use acceptable method for contraception for duration of study.
* Histologically-confirmed indolent or mantle cell lymphoma, utilizing the World Health Organization (WHO) classification. The biopsy must fulfill one of the following criteria:

  * Follicular lymphoma, grades 1-3
  * Marginal zone lymphoma
  * Small lymphocytic lymphoma (circulating lymphocyte count must be < 5,000)
  * Lymphoplasmacytic lymphoma
  * Mantle cell lymphoma [confirmed by cyclin D1+ or FISH for t(11;14)]
* Age ≥ 18 years
* Must have received at least one prior chemotherapy regimen for lymphoma. Patients treated only with antibody therapy or only with radiation therapy are not eligible.
* Zubrod performance status ≤ 3
* Patients must have measurable disease or an indication to receive additional therapy

Exclusion Criteria:

* Patient has platelet count of ≤75,000/mm^3 within 14 days before enrollment.
* Patient has absolute neutrophil count of < 1,000/mm^3 within 14 days before enrollment.
* Patient has calculated or measured creatinine clearance of <30 mL/minute within 14 days before enrollment.
* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to boron or mannitol
* Female subject is pregnant or breast-feeding. Confirmation subject is not pregnant must be established by negative serum ß-human chorionic gonadotropin (ß-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received chemotherapy or antibody therapy within 28 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patient has received other investigational drugs with 14 days before enrollment
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Prior exposure to bendamustine
* Prior exposure to bortezomib if Time to Progression (TTP) after bortezomib containing regimen was < 6 months. If TTP after bortezomib containing regimen was > 6 months, then patient is allowed to enroll on the study.
* Patient has concomitant active malignancy requiring therapy
* Patient is known to be HIV positive (test result not required for enrollment).
* History of solid organ transplantation, or post transplant lymphoproliferative disorder
* Patient has history of allogeneic stem cell transplantation.
* Patient has history of autologous stem cell transplantation or radioimmunotherapy within the previous 4 months.
* Patient has received any other investigational drugs within 14 days prior to enrollment
* History of, or clinically apparent CNS lymphoma
* Any clinically significant abnormality in screening blood chemistry, hematology, or urinalysis results that, in the judgment of the investigator, would impede adequate evaluation of adverse events and/or response to treatment, or that requires aggressive intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Friedberg, md, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - Nebraska Medical Center, Omaha, Nebraska
  - Cornell Wiell Medical College, New York, New York
  - University of Rochester Medical Center (James P. Wilmot Cancer Center), Rochester, New York

REFERENCES:
- [Derived] Friedberg JW, Vose JM, Kelly JL, Young F, Bernstein SH, Peterson D, Rich L, Blumel S, Proia NK, Liesveld J, Fisher RI, Armitage JO, Grant S, Leonard JP. The combination of bendamustine, bortezomib, and rituximab for patients with relapsed/refractory indolent and mantle cell non-Hodgkin lymphoma. Blood. 2011 Mar 10;117(10):2807-12. doi: 10.1182/blood-2010-11-314708. Epub 2011 Jan 14. PMID 21239695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at the University of Rochester Medical Center, Weill Cornell Medical Center and the University of Nebraska began in October 2007 and ended in March 2009. Patients were recruited in a medial clinic setting.
Groups:
- Lymphoma Subjects: Subjects that met all eligibility criteria and were given study treatment.
Period: Overall Study
Arm/Group | Lymphoma Subjects
Started | 30 (31 patients enrolled; one patient was determined to be ineligible, and did not receive any therapy.)
Completed | 19 (25 patients received at least 4 cycles. 29 patients were evaluable for response.)
Not Completed | 11
Not completed — Adverse Event | 7
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lymphoma Subjects
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival at 2 Years
Description: To determine the progression-free survival following treatment with the BVR combination in patients with relapsed or refractory indolent and mantle cell non-Hodgkin lymphoma.
Time Frame: Two years
Population: Analysis was per protocol.
Measure: Number; unit: Participants
Groups:
- Lymphoma Subjects: Subjects that met all eligibility criteria and were treated.
Arm/Group | Lymphoma Subjects
Number analyzed (Participants) | 29
Participants | 13

2. Secondary Outcome: Toxicity of Drug Combination in the Subjects
Time Frame: Two years
Measure: Number; unit: Lymphoma Subjects
Arm/Group | Lymphoma Subjects
Number analyzed (Participants) | 29
Lymphoma Subjects | 13

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR)to protocol treatment - Partial response, Complete response, etc.
Time Frame: Two years
Measure: Number; unit: Lymphoma Subjects
Arm/Group | Lymphoma Subjects
Number analyzed (Participants) | 29
Lymphoma Subjects | 13

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Lymphoma Subjects
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphoma Subjects (N=30)
Sepsis (Gastrointestinal disorders) | 1 (1)
Liver Failure (Gastrointestinal disorders) | 1 (1)
Renal Failure (Endocrine disorders) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Hypotension (Blood and lymphatic system disorders) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphoma Subjects (N=30)
Nausea (Gastrointestinal disorders) | 15 (15)
Peripheral neuropathy (Nervous system disorders) | 14 (14)
Fatigue (General disorders) | 14 (14)
Constipation (Gastrointestinal disorders) | 12 (12)
Fever (General disorders) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Cough (Infections and infestations) | 7 (7)
Hypotension (Cardiac disorders) | 6 (6)
Rigors / chills (General disorders) | 5 (5)
Pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Herpes zoster (Infections and infestations) | 4 (4)
Allergic reaction (Infections and infestations) | 4 (4)
Headache (General disorders) | 4 (4)
Pruritis (General disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 3 (3)
Dizziness (General disorders) | 3 (3)
Rash (Infections and infestations) | 3 (3)
Shortness of breath (Cardiac disorders) | 3 (3)
Stomach/abdominal pain (Gastrointestinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
19 patients received a full 6 cycles of therapy. All patients received at least one cycle of therapy, 25 patients received at least 4 cycles. Reasons for early termination included progressive disease and toxicity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes